CLINICAL TRIAL: NCT02321072
Title: The Effects of Hyperoxia on Organ Dysfunction and Outcome in Critically Ill Patients With SIRS
Brief Title: Optimal Oxygenation in the Intensive Care Unit
Acronym: O2-ICU
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Tergooi Hospital (Other)
Responsible Party: Principal Investigator, Angelique Spoelstra-de Man, Consultant Intensivist, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2014/459; 2014-003468-19 (EudraCT Number)
Record Dates: First submitted 2014-12-09; First posted 2014-12-22 (Estimated); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Systemic Inflammatory Response Syndrome
Keywords: oxygen; hypoxia; hyperoxia; critical care; intensive care
MeSH Terms: conditions — Systemic Inflammatory Response Syndrome; Hypoxia; Hyperoxia | interventions — Oxygen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High-normal PaO2 (Active Comparator): In patients requiring respiratory monitoring, supplemental oxygen is titrated to achieve a PaO2 of 120 mmHg (16 kPa), range 105-135 mmHg (14-18 kPa).
  Interventions: Drug: Oxygen
- Low-normal PaO2 (Active Comparator): In patients requiring respiratory monitoring, supplemental oxygen is titrated to achieve a target PaO2 of 75 mmHg (10 kPa), range 60-90 mmHg (8-18 kPa).
  Interventions: Drug: Oxygen

INTERVENTIONS:
Drug: Oxygen

SUMMARY:
Objectives:

1. To study the short- and long-term effect of two different PaO2 targets on circulatory status, organ dysfunction and outcome in patient admitted to the ICU with Systemic Inflammatory Response Syndrome (SIRS) criteria.
2. To study underlying mechanisms of hyperoxia by determining differences in oxidative stress response between the hyperoxic and the normoxic patients.

Study design:

Randomized, prospective multicentre clinical trial

Study population:

Patients admitted to the Intensive Care unit with ≥ 2 positive SIRS-criteria and an expected ICU stay of more than 48 hours

Intervention:

Group 1: target PaO2 120 (105 - 135) mmHg (high-normal)

Group 2: target PaO2 75 (60 - 90) mmHg (low-normal)

Primary endpoints:

The primary endpoint will be cumulative daily delta SOFA score (CDDS) from day 1 to day 14.

DETAILED DESCRIPTION:
Rationale:

Contrary to hypoxia, many physicians do not consider hyperoxia harmful for their patients. To prevent hypoxia, superfluous administration of oxygen is common practice, and hyperoxia is seen in many patients, especially on Intensive Care units. However, an increasing number of studies not only confirm the known negative pulmonary effects of chronic oxygen oversupply, but also important and more acute circulatory effects, characterised by decreased cardiac output (CO), increased systemic vascular resistance (SVR), and impaired microvascular perfusion. These phenomena can impair perfusion of organs, which may outweigh higher arterial oxygen content, resulting in a net loss of oxygen delivery and perturbed organ function. This may for example be responsible for hyperoxia-associated increased infarct size and increased mortality after myocardial infarction and cardiac arrest. The underlying mechanisms are not clarified yet, but probably involve increased oxidative stress with systemic vasoconstriction.

On the other hand, hyperoxia can also induce several favourable effects. The majority of ICU-patients have a systemic inflammatory response syndrome (SIRS) with concomitant vasoplegia due to trauma, sepsis or ischemia/reperfusion injury. Vasoconstriction could benefit these patients with severe SIRS, reducing the need for intravenous volume resuscitation and vasopressor requirements. Furthermore, hyperoxia may exert a preconditioning effect in patients with ischemia/reperfusion injury and prevent new infections due to its antibacterial properties.

Hypothesis:

Hyperoxia during SIRS ultimately has unfavourable effects on organ function, especially on a longer term.

Objectives:

1. To study the short- and long-term effect of two different PaO2 targets on circulatory status, organ dysfunction and outcome.
2. To study underlying mechanisms of hyperoxia by determining differences in oxidative stress response between the hyperoxic and the normoxic patients.

Study design:

Randomized, prospective multicentre clinical trial

Study population:

Patients admitted to the Intensive Care unit with ≥ 2 positive SIRS-criteria and an expected ICU stay of more than 48 hours

Intervention:

We will investigate 2 groups with PaO2 targets both within the range of current practice

Group 1: target PaO2 120 (105 - 135) mmHg (high-normal)

Group 2: target PaO2 75 (60 - 90) mmHg (low-normal)

ELIGIBILITY:
Inclusion Criteria:

* ≥2 positive SIRS-criteria:

  * Temperature >38 deg.C or hypothermia <36 deg.C
  * Heart rate >90 bpm
  * Respiratory rate >20 /min or pCO2 <32 mmHg (4.3 kPa)
  * Number of leucocytes >12 x 10^9/l of <4 x 10^9/l of >10% bands
* Within 12 hours of admittance to the ICU
* Expected stay of more than 48 hours as estimated by the attending physician

Exclusion Criteria:

* Elective surgery
* Carbon monoxide poisoning
* Cyanide intoxication
* Methemoglobinemia
* Sickle cell anemia
* Severe pulmonary arterial hypertension (WHO class III or IV)
* Known severe Acute Respiratory Distress Syndrome (ARDS) (PaO2/FiO2 ≤100 mmHg and PEEP ≥ 5 cm H2O)
* Known cardiac right to left shunting
* Pregnancy
* Severe Chronic Obstructive Pulmonary Disease (COPD) (Gold class III or IV) or other severe chronic pulmonary disease
* Patients participating in other interventional trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Daily Delta Sequential Organ Failure Assessment Score | 14 days
  The primary endpoint will be cumulative daily delta SOFA score (CDDS) from day 1 to day 14, calculated as the sum of [daily SOFA score minus admission SOFA score] from day 2 to day 14.
  Daily SOFA score is calculated as the total of maximum scores for each organ system excluding respiratory system (because of possible PaO2/FiO2 distortion). For patients discharged from the ICU, SOFA score will be registered as 0 from the day of discharge to day 14. Death in the ICU will be registered as a score of 20 (maximum) from the day of death to day 14.

SECONDARY OUTCOMES:
total maximum SOFA score minus SOFA score on admission | 14 days
SOFA rate of decline | 14 days
Total maximum SOFA score, total maximum SOFA score minus SOFA score on admission, SOFA rate of decline | 14 days
Mortality | 14 days, in-ICU (max 90 days), in-hospital (max 90 days)
Hypoxic events (PaO2 <55 mmHg) | 14 days
Vasopressor / Inotrope requirements | 14 days
Renal function, fluid balance | 14 days
Oxidative stress (F2-isoprostanes) | days 1, 3, 7
Duration of mechanical ventilation and ventilator-free days | 14 days
Length of stay (ICU) | average expected 2 to 28 days
Length of stay (hospital) | average expected 10 to 28 days
Systemic Vascular Resistance Index | 14 days
  In a random subpopulation.
Cardiac Index | 14 days
  In a random subpopulation.
Microcirculatory flow index and Perfused vessel density | 14 days
  In a random subpopulation. Composite endpoint for two sidestream dark-field microcirculatory measurements.

CONTACTS AND LOCATIONS:
Overall Officials: A.M.E. de Man, MD, PhD, Principal Investigator — Amsterdam UMC, location VUmc
Locations (1):
- VU University Medical Center, Amsterdam, Netherlands

REFERENCES:
- [Derived] Klitgaard TL, Schjorring OL, Nielsen FM, Meyhoff CS, Perner A, Wetterslev J, Rasmussen BS, Barbateskovic M. Higher versus lower fractions of inspired oxygen or targets of arterial oxygenation for adults admitted to the intensive care unit. Cochrane Database Syst Rev. 2023 Sep 13;9(9):CD012631. doi: 10.1002/14651858.CD012631.pub3. PMID 37700687
- [Derived] Gelissen H, de Grooth HJ, Smulders Y, Wils EJ, de Ruijter W, Vink R, Smit B, Rottgering J, Atmowihardjo L, Girbes A, Elbers P, Tuinman PR, Oudemans-van Straaten H, de Man A. Effect of Low-Normal vs High-Normal Oxygenation Targets on Organ Dysfunction in Critically Ill Patients: A Randomized Clinical Trial. JAMA. 2021 Sep 14;326(10):940-948. doi: 10.1001/jama.2021.13011. PMID 34463696